CLINICAL TRIAL: NCT04119739
Title: Pain Reduction Produced by Physiotherapy, Ibuprofen Arginine, and the Absence of Treatment, in Carpal Tunnel Syndrome
Brief Title: Pain Reduction Produced by Different Treatments in Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Francisco Unda Solano (Other)
Responsible Party: Sponsor-Investigator, Francisco Unda Solano, Biomedicine Doctorate Program Investigator, Universidad Europea de Madrid
Organization: Universidad Europea de Madrid (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CE0072015-02-02
Record Dates: First submitted 2019-10-06; First posted 2019-10-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Ibuprofen; Median nerve neural mobilization; Waiting list control group; Physiotherapy; Pain management
MeSH Terms: conditions — Carpal Tunnel Syndrome; Agnosia | interventions — ibuprofen arginine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Median nerve neural mobilization (Experimental): Non pharmaceutical, non invasive, physiotherapy technique; which consists of a passive and repetitive upper limb movement that seeks to induced median nerve gliding and incursions against surrounding connective tissue. Subjects will be treated 5 days per week during a total time lapse of 4 weeks.
  Interventions: Other: Median nerve neural mobilization
- Ibuprofen Arginine (Active Comparator): Oral tablet pharmaceutical treatment. Participants will be treated with a maximum of 1200 mg per day, subdivided in 3 intakes of 400 mg each 8 hours during a time lapse of 4 weeks.
  Interventions: Drug: Ibuprofen Arginine
- Control group (No Intervention): Waiting list control group. Participants that belong to the no intervention arm will be assigned to a waiting list to receive treatment. The participants will not receive treatment for carpal tunnel syndrome during a time lapse of 4 weeks. After this period of time, participants will begin the best treatment available.

INTERVENTIONS:
Other: Median nerve neural mobilization — Manual therapy maneuver performed in the upper limb.
  Arms: Median nerve neural mobilization
Drug: Ibuprofen Arginine — Oral tablets
  Other Names: Spedifen; FASPIC
  Arms: Ibuprofen Arginine

SUMMARY:
Pain reduction effects of the median nerve neural mobilization technique (a physiotherapy treatment) will be compared to those produced by a pharmaceutical treatment and the absence of treatment, in subjects who suffer carpal tunnel syndrome.

DETAILED DESCRIPTION:
The present randomized clinical trial will perform a comparison of the pain reduction effects produced by the application of median nerve neural mobilization (non invasive and non pharmaceutical physiotherapy treatment), to the pain reduction effect produced by an oral ibuprofen treatment or the lack of treatment (waiting list control group) in subjects diagnosed with carpal tunnel syndrome. Additionally, effects over the functionality of the affected upper limb will be evaluated and compared. Subjects will be invited to participate and randomly allocated to 3 different groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be medically diagnosed with unilateral carpal tunnel syndrome (with confirmative electrodiagnostic findings).
* Full understanding of written and spoken Spanish (language).
* Participants must freely consent to participate.
* The presence of positive Phalen and Tinel signs.
* The presence of carpal tunnel syndrome signs and symptoms

Exclusion Criteria:

* The lack to meet inclusion criterions, the presence of cognitive impairment.

  * Tumors
  * Cancer
  * Upper limb surgery or trauma
  * Pregnancy
  * Deformities of the (affected) upper limb
  * Recent skin injuries or infections (in the affected upper limb)
  * Autoimmune inflammatory conditions or flu type symptoms.
  * Allergy to gabapentin, ibuprofen or ibuprofen arginine
  * Participants must not be (during the present investigation) under any type of pain reducing treatment (conservative, homeopathic, invasive or not invasive).
  * Metabolic neuropathy.
  * Obesity (body mass index over 30).
  * Participants who are not employed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Distal upper limb pain | Changes from baseline (measured immediately before the application of the first treatment) and 40 minutes after the application of the last treatment.
  Assessed through the visual analog scale (VAS). The VAS is a psychometric response scale. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.The VAS is the most frequently used method to assess pain intensity. The scale will be displayed as a horizontal 10-cm line labelled at each end by descriptors such as 'no pain' (the minimum and best outcome possible) and 'worse pain ever' (maximum and worst outcome possible). The participant will mark the line to indicate pain severity and it is simply quantified by measuring the distance in centimeters from 0 (no pain) to the patient's marked rating.

SECONDARY OUTCOMES:
Upper limb function | Changes from baseline (measured immediately before the application of the first treatment) and at 40 minutes after the application of the last treatment.
  Assessed through the Quick- Disabilities of the Arm, Shoulder and Hand (Quick- DASH) questionary, which is a shortened version of the 30-item Disabilities of the Arm, Shoulder and Hand (DASH) instrument. The instrument administered to the participants will be a self-report questionnaire, that will rate the difficulty and interference of daily life on a 5 point Likert scale. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability).

OTHER OUTCOMES:
Work Status at baseline | Measured immediately before the application of the first treatment
  This measure is performed through the employed participant (full-time or part-time) answering in a dichotomous manner (yes or no) the question: "Do you currently work?"
Work Status post treatment | Measured immediatly after the application of the last treatment.
  This measure is performed through the employed participant (full-time or part-time) answering in a dichotomous manner (yes or no) the question: "Do you currently work?"
Change in Work Task (Job Type) | Measured immediatly after the application of the last treatment.
  This measure is performed through the employed participant (full-time or part-time) answering in a dichotomous manner (yes or no) the question: "Did you change your job type or task?"
Tampa Scale for Kinesiophobia-17 (TSK-17 | Changes from baseline (measured immediately before the application of the first treatment), and at 60 minutes after the application of the last treatment.
  The Tampa Scale for Kinesiophobia-17 (TSK-17) is a 17-item questionnaire designed to assess the fear of movement and re-injury (kinesiophobia). Items are rated on a 4-point Likert scale (ranging from "strongly disagree" to "strongly agree"), yielding a total score that reflects the severity of pain-related fear avoidance beliefs. It's a widely used and vailidaded clinical and research instrument. The standard total score range for the Tampa Scale for Kinesiophobia (TSK-17) is 17 to 68. It is calculated by summing 17 items, each scored 1-4, with four items reverse-scored. Higher scores indicate greater fear of movement.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Unda Solano, PHD, Principal Investigator
Locations (1):
- Ciudad Hospitalaria Enrique Tejera, Valencia, Carabobo, Venezuela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ilyas AM, Miller AJ, Graham JG, Matzon JL. A Prospective, Randomized, Double-Blinded Trial Comparing Acetaminophen, Ibuprofen, and Oxycodone for Pain Management After Hand Surgery. Orthopedics. 2019 Mar 1;42(2):110-115. doi: 10.3928/01477447-20190221-02. Epub 2019 Feb 27. PMID 30810754
- [Background] Choi GH, Wieland LS, Lee H, Sim H, Lee MS, Shin BC. Acupuncture and related interventions for the treatment of symptoms associated with carpal tunnel syndrome. Cochrane Database Syst Rev. 2018 Dec 2;12(12):CD011215. doi: 10.1002/14651858.CD011215.pub2. PMID 30521680
- [Background] Weinheimer K, Michelotti B, Silver J, Taylor K, Payatakes A. A Prospective, Randomized, Double-Blinded Controlled Trial Comparing Ibuprofen and Acetaminophen Versus Hydrocodone and Acetaminophen for Soft Tissue Hand Procedures. J Hand Surg Am. 2019 May;44(5):387-393. doi: 10.1016/j.jhsa.2018.10.014. Epub 2018 Nov 27. PMID 30502019
- [Background] Riasi H, Rajabpour Sanati A, Salehi F, Salehian H, Ghaemi K. Analyzing the therapeutic effects of short wrist splint in patients with carpal tunnel syndrome (CTS) under ibuprofen treatment from an EMG-NCV perspective. J Med Life. 2015;8(Spec Iss 4):154-158. PMID 28316723
- [Background] Davis PT, Hulbert JR, Kassak KM, Meyer JJ. Comparative efficacy of conservative medical and chiropractic treatments for carpal tunnel syndrome: a randomized clinical trail. J Manipulative Physiol Ther. 1998 Jun;21(5):317-26. PMID 9627862
- [Background] Sanz DR, Solano FU, Lopez DL, Corbalan IS, Morales CR, Lobo CC. Effectiveness of median nerve neural mobilization versus oral ibuprofen treatment in subjects who suffer from cervicobrachial pain: a randomized clinical trial. Arch Med Sci. 2018 Jun;14(4):871-879. doi: 10.5114/aoms.2017.70328. Epub 2017 Sep 26. PMID 30002707
- [Background] Calvo-Lobo C, Unda-Solano F, Lopez-Lopez D, Sanz-Corbalan I, Romero-Morales C, Palomo-Lopez P, Seco-Calvo J, Rodriguez-Sanz D. Is pharmacologic treatment better than neural mobilization for cervicobrachial pain? A randomized clinical trial. Int J Med Sci. 2018 Mar 8;15(5):456-465. doi: 10.7150/ijms.23525. eCollection 2018. PMID 29559834
- [Background] Rodriguez-Sanz D, Lopez-Lopez D, Unda-Solano F, Romero-Morales C, Sanz-Corbalan I, Beltran-Alacreu H, Calvo-Lobo C. Effects of Median Nerve Neural Mobilization in Treating Cervicobrachial Pain: A Randomized Waiting List-Controlled Clinical Trial. Pain Pract. 2018 Apr;18(4):431-442. doi: 10.1111/papr.12614. Epub 2017 Nov 20. PMID 28734105
- [Background] Basson A, Olivier B, Ellis R, Coppieters M, Stewart A, Mudzi W. The Effectiveness of Neural Mobilization for Neuromusculoskeletal Conditions: A Systematic Review and Meta-analysis. J Orthop Sports Phys Ther. 2017 Sep;47(9):593-615. doi: 10.2519/jospt.2017.7117. Epub 2017 Jul 13. PMID 28704626
- [Background] Ballestero-Perez R, Plaza-Manzano G, Urraca-Gesto A, Romo-Romo F, Atin-Arratibel MLA, Pecos-Martin D, Gallego-Izquierdo T, Romero-Franco N. Effectiveness of Nerve Gliding Exercises on Carpal Tunnel Syndrome: A Systematic Review. J Manipulative Physiol Ther. 2017 Jan;40(1):50-59. doi: 10.1016/j.jmpt.2016.10.004. Epub 2016 Nov 11. PMID 27842937
- [Background] Shin D, Lee SJ, Ha YM, Choi YS, Kim JW, Park SR, Park MK. Pharmacokinetic and pharmacodynamic evaluation according to absorption differences in three formulations of ibuprofen. Drug Des Devel Ther. 2017 Jan 4;11:135-141. doi: 10.2147/DDDT.S121633. eCollection 2017. PMID 28115830
- [Background] Eren Y, Yavasoglu NG, Comoglu SS. The relationship between QDASH scale and clinical, electrophysiological findings in carpal tunnel syndrome. Adv Clin Exp Med. 2018 Jan;27(1):71-75. doi: 10.17219/acem/67947. PMID 29521045